CLINICAL TRIAL: NCT02025816
Title: RNAseq Analysis of Microbial Gene Expression in Necrotizing Soft Tissue Infections
Acronym: NSTI
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor
Other Study IDs: L14-002
Record Dates: First submitted 2013-12-30; First posted 2014-01-01 (Estimated); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Necrotizing Soft Tissue Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Tissue biopsies for RNAseq analysis of microbial gene expression
Oversight: Data Monitoring Committee: No

SUMMARY:
Hypothesis: We hypothesize that RNAseq will allow us to learn more about the causative agents of necrotizing soft tissue infections (NSTI) and risk factors involved in acquiring these devastating infections

Tissue biopsies will be obtained from consented patients admitted with NSTI. Biopsies will be used for standard clinical analysis of bacterial species present or stored for later RNA sequencing. RNA sequencing will identify bacteria that are present within the infection site that may not be detected using standard culture techniques as well as reveal bacterial gene expression profiles within the NSTI site. Medical charts will also be reviewed for basic patient information as well as wound care management practices. We hope to identify bacterial species commonly present in these types of infections as well as risk factors predisposing individuals to NSTI's.

ELIGIBILITY:
Inclusion Criteria:

* Patient or LAR agrees to the procedure and signs informed consent form
* Patient is at least 18 yrs of age
* Patient has been diagnosed with an NSTI

Exclusion Criteria:

* Patient not willing to undergo additional tissue biopsies for RNA sequencing analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Twenty to twenty five patients with necrotizing soft tissue infections (NSTI) admitted to the University Medical Center, Lubbock, TX
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with non-culturable, anaerobic bacterial species colonization of NSTI | 2-6 wks (duration of hospitalization)

CONTACTS AND LOCATIONS:
Overall Officials: Kendra Rumbaugh, PhD, Principal Investigator — Texas Tech University Health Sciences Center
Locations (2):
- United States (2):
  - Texas Tech University Health Sciences Center/University Medical Center, Lubbock, Texas
  - University Medical Center, Lubbock, Texas